CLINICAL TRIAL: NCT02832310
Title: The Effects of Valsalva Maneuver on Head, Neck and Upper Extremity Arterial Systems
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, fatih altıparmak, Resident, Tokat Gaziosmanpasa University
Other Study IDs: 16-KAEK-037
Record Dates: First submitted 2016-03-30; First posted 2016-07-14 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Asymptomatic Diseases
Keywords: valsalva
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Valsalva Maneuver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: valsalva maneuver — the effects of valsalva maneuver on arterial pressure

SUMMARY:
The aim of this study is to determine the relation between arterial diameter and flow of carotis interna, brachial artery and radial artery before and after valsalva maneuver.

DETAILED DESCRIPTION:
The aim of this study is to determine the relation between arterial diameter and flow of carotis interna, brachial artery and radial artery before and after valsalva maneuver. A total of 70 patients in preoperative period will enroll in this study. After a deep inspiration, patients will asked to exhale to a valf system with a flow pressure of 20-40 mmHg and duration of 15 seconds. During valsalva maneuver, the diameter and flow rates of carotis interna, brachial artery and radial artery will measure using ultrasound. All data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists score of I, II, III

Exclusion Criteria:

* Morbid obesity (body mass index over 40)
* Not to participate in the study
* Psychiatric diseases
* Peripheral vascular diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: peroperative patients, healhty volunteers
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
arterial flow rate | 1 year

SECONDARY OUTCOMES:
arterial diameter | 1 year

IPD SHARING:
Plan to Share IPD: No